CLINICAL TRIAL: NCT04465162
Title: Radiation Therapy Alone for Stage 1 and 2 MALT (Mucosa-Associated Lymphoid Tissue) Lymphoma
Brief Title: Radiation Therapy Alone for the Treatment of Stage 1 and 2 Mucosa-Associated Lymphoid Tissue (MALT) Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID99-384; NCI-2020-02549 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ID99-384 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-05-06; First posted 2020-07-09 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Ann Arbor Stage I Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Ann Arbor Stage II Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Extranodal Marginal Zone Lymphoma
MeSH Terms: interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy) (Experimental): Patients undergo radiation therapy QD 5 times weekly over 3.5-5 weeks.
  Interventions: Other: Radiation Therapy

INTERVENTIONS:
Other: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This trial studies the side effects of radiation therapy used alone, and if it can achieve a high cure rate in the treatment of patients with MALT lymphoma. Radiation therapy uses high energy sources to kill cancer cells and shrink tumors. This treatment may improve the patient's lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy and toxicity of radiation therapy alone in treating stage 1 and 2 MALT lymphoma for newly diagnosed patients and for the patients who failed other treatment modalities.

OUTLINE:

Patients undergo radiation therapy once daily (QD) 5 times weekly over 3.5-5 weeks.

After completion of study treatment, patients are followed up at 6-8 weeks, and then every 3-4 months for year 1, every 4-6 months for year 2, every 6 months for years 3 and 4, and once yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stage 1 and 2 MALT lymphoma are eligible for this study
* Patients with Helicobacter (H.) pylori positive gastric MALT lymphoma are recommended to have treatments with antibiotics prior to enrollment to this protocol
* Patients who failed other treatment modalities (e.g. chemotherapy, antibiotics therapy etc) are also eligible as far as they never had stage 3 or 4 disease during the course of the disease or disease progression to the opposite side of the diaphragm (as the time course of the response to antibiotic therapy can be very variable among patients, sometimes requiring more than one year for complete response, failure to antibiotic therapy can be very variable among patients, sometimes requiring more than one year for complete response, failure to antibiotic treatment will be defined as no response or progression of the disease documented by endoscopy and biopsy)
* Patients who have had stage 4 diseases due to bilateral parotid gland or ocular/ocular adnexal involvement or due to multiple sites within Waldeyer's ring will still be eligible

Exclusion Criteria:

* Patients who had previous radiation dose to the site of the current primary disease which would lead to violation of known radiation tolerance limit of that particular site if treated again
* Patients with MALT lymphoma of the skin whose lesions are separated by more than 5 cm will be ineligible
* Previous or concurrent malignancy in any form would not be an exclusion criterion. However, patients who receive chemotherapy for concurrent malignancy will be excluded from statistical analysis
* Low blood cell counts would not be exclusion criteria as far as the patient is willing to accept supportive measures such as transfusions, filgrastim and epoetin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2000-06-07 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina S Dabaja, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Fang P, Gunther JR, Pinnix CC, Dong W, Strati P, Nastoupil LJ, Steiner RE, Ahmed S, Damron EP, Fowler N, Nair R, Westin JR, Neelapu S, Ha CS, Dabaja BS. A Prospective Trial of Radiation Therapy Efficacy and Toxicity for Localized Mucosa-associated Lymphoid Tissue (MALT) Lymphoma. Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1414-1420. doi: 10.1016/j.ijrobp.2020.11.070. Epub 2020 Dec 10. PMID 33309978
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 75 participants enrolled in study, 2 participants did not receive Radiation Therapy(RT); 1 owing to discovered stage III disease and 1 who chose observation after complete surgical resection of disease in a gastric polyp.
Period: Overall Study
Arm/Group | Treatment (Radiation Therapy)
Started | 73
Completed | 73
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 73
Age, Continuous [Median (Full Range); unit: years] | 57 [25 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 73
Clinical Stage [Count of Participants; unit: Participants] — Stage I. This stage is usually a cancer that has not grown deeply into nearby tissues. It also has not spread to the lymph nodes or other parts of the body. It is often called early-stage cancer. Stage II and Stage III. In general, these 2 stages are cancers that have grown more deeply into nearby tissue. They may have also spread to lymph nodes but not to other parts of the body. Stage IV. This stage means that the cancer has spread to other organs or parts of the body. It may be also called advanced or metastatic cancer.
  Participants
    I | 61
    II | 10
    IV | 2
Tumor Location [Count of Participants; unit: Participants]
  Head and neck (nonorbit) | 13
  Orbit | 17
  Stomach | 34
  Skin | 4
  Other | 5
Helicobacter pylori positive at initial diagnosis [Count of Participants; unit: Participants] — Population: Participants with gastric Mucosa-Associated Lymphoid Tissue (MALT) and were Helicobacter pylori positive at the time of initial diagnosis.
  Participants
    number analyzed (Participants) | 34
    (all) | 13
Treatment before radiation therapy [Count of Participants; unit: Participants]
  Antibiotics | 22
  Rituximab | 3
  Surgery | 19
  Other | 1
  None | 27
  Unknown | 1
Radiation dose, Gy [Count of Participants; unit: Participants]
  24-28.5 | 8
  30-30.6 | 45
  33-39.6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival (RFS)
Description: RFS was defined as the time in months from the date of study entry until the last follow-up or death, with all deaths censored. Kaplan-Meier curves were estimated for the survival distributions.
Time Frame: Through study completion, up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 73
months | 83 [74 to 93]

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to progression or death. Kaplan-Meier curves were estimated for the survival distributions.
Time Frame: 17.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 73
months | 17.5 [11.5 to NA] — survival curve for upper limit does not cross 50% survival

3. Secondary Outcome: Progression Free Survival (PFS) at 10 Years
Description: PFS events is the time in months and defined as any lymphoma relapse ( lymphoma that comes back after successful treatment and a period of remission) or death from any cause. Kaplan-Meier curves were estimated for the survival distributions.
Time Frame: Through study completion, up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 73
months | 73 [60 to 84]

4. Secondary Outcome: 10 Year Overall Survival (OS)
Description: Overall Survival is the time in months from start of study treatment to date of death due to any cause. Overall survival rates are estimated by the Kaplan-Meier method.
Time Frame: Through study completion, up to 10 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Radiation Therapy)
Number analyzed (Participants) | 73
months | 86 [77 to 96]

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study medication, All-Cause Mortality was assessed up to 10 years, and Serious and Other (Not Including Serious) adverse events were assessed up to 9 weeks
Arm/Group | Treatment (Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 11/73
Serious Adverse Events (participants affected / at risk) | 0/73
Other Adverse Events (participants affected / at risk) | 28/73
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Radiation Therapy) (N=73)
Fatigue (Gastrointestinal disorders) | 13
Dermatitis (Skin and subcutaneous tissue disorders) | 24
Eye toxicities (Eye disorders) | 13
Erythema (Skin and subcutaneous tissue disorders) | 1
Retinopathy (Eye disorders) | 1
Cataracts (Eye disorders) | 6
Xerostomia (Eye disorders) | 7
Ear (Ear and labyrinth disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Skin (Skin and subcutaneous tissue disorders) | 24
Larynx (Respiratory, thoracic and mediastinal disorders) | 5
Salivary (Gastrointestinal disorders) | 8
Mucositis (Respiratory, thoracic and mediastinal disorders) | 5
Pharynx (Respiratory, thoracic and mediastinal disorders) | 12
Upper GI (Gastrointestinal disorders) | 28
Lower GI (Gastrointestinal disorders) | 5
Genitourinary (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Lung (Respiratory, thoracic and mediastinal disorders) | 1
Bone (General disorders) | 1
Bladder (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT04465162/Prot_SAP_000.pdf